CLINICAL TRIAL: NCT06010290
Title: The Novel 18F-labeled MAO-B PET/CT Imaging on Parkinsonism Patients of Chinese Population: a Prospective Study
Brief Title: The Novel 18F-labeled MAO-B PET Tracer Study in Parkinsonism Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: MAO-B PET/CT STUDY
Record Dates: First submitted 2023-08-10; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2022-11

CONDITIONS: Parkinson Disease
Keywords: PET/CT
MeSH Terms: conditions — Parkinson Disease | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinsonism patients: This group/cohort comprises clinically diagnosed as Parkinsonism, including Parkinson's disease and atypical Parkinsonism syndromes, and each participant is injected 18F-SMBT-1 (185-370Mbq) and underwent PET/CT scanning within 50-70 min after injection.
  Interventions: Drug: 18F-SMBT-1
- Health control: Each participant is injected 18F-SMBT-1 (185-370Mbq) and underwent PET/CT scanning within 50-70 min after injection.
  Interventions: Drug: 18F-SMBT-1

INTERVENTIONS:
Drug: 18F-SMBT-1 — Each participant receives intravenous injection of 18F-SMBT-1, and undergo PET/CT imaging within the special time. 18F-FP-CIT and 18F-FDG PET/CT are used to assess the change of cerebral dopamine transporters and glucose metabolism for auxiliary diagnosis.
  Other Names: 18F-FP-CIT; 18F-FDG

SUMMARY:
This study mainly aims to prospectively evaluate the changes of reactive astrogliosis in Parkinsonism patients of Chinese population by the novel 18F-labeled MAO-B PET tracer.

DETAILED DESCRIPTION:
18F-SMBT-1, the novel 18F-labeled MAO-B PET tracer, was evaluated reactive astrogliosis in Alzheimer's disease successfully. In this prospective study, we assess the changes of reactive astrocytes in cerebral gray matter and white matter on Parkinson's disease by 18F-SMBT-1 PET/CT imaging among Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 40 to 90 years old.
* Clinically diagnosed as Parkinsonism, including Parkinson's disease and atypical Parkinsonism syndromes.
* Can cooperate with 18F-FDG PET/CT, 18F-FP-CIT PET/CT and 3D T1-weighted structural MR scans.
* Complete clinical data, including modified Hoehn and Yahr staging scale and the Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS).

Exclusion Criteria:

* Cannot cooperate with PET/CT or MR examination.
* Associated with brain diseases such as stroke, brain trauma, brain tumor, and cranial surgery.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population are recruited from the Department of Neurology of the First Affiliated Hospital of University of Science and Technology of China (USTC).
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Standard uptake value ratio (SUVR) | 60 days
  Standard uptake value ratio of 18F-SMBT-1, 18F-FP-CIT and 18F-FDG in the key cerebral regions using the cerebellar cortex or subcortical white matter as a reference region
Clinical parameters | 60 days
  Clinical parameters include sex, age, Hoehn-Yahr Stage, and Unified Parkinson's disease rating scale (UPDRS).

SECONDARY OUTCOMES:
Correlation coefficient 1 | 60 days
  Correlation analysis of SUVR between 18F-SMBT-1, 18F-FP-CIT and 18F-FDG in the key cerebral regions.
Correlation coefficient 2 | 60 days
  Correlation analysis between SUVR of 18F-SMBT-1 PET/CT in the key cerebral regions and clinical parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Xie, MD, Study Chair — The First Affiliated Hospital of China University of Science and Technology
Locations (1):
- The First Affiliated Hospital of China University of Science and Technology, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No